CLINICAL TRIAL: NCT01404221
Title: The Combination of Biochemical Markers and Two and Three Dimensional Ultrasound Using Geometric Morphometrics in the Identification of Congenital Anomalies and Maternal or Fetal Complications
Brief Title: Biochemical Markers and 2 and 3D Ultrasound to ID Maternal & Fetal Complications
Status: Terminated | Type: Observational
Why Stopped: No safety issues. Need to rewrite protocol
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Burt Rochelson, Investigator, MD, Northwell Health
Other Study IDs: IRB 07-077
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Pregnancy; Fetal Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Can a combination of prenatal screening blood tests, early ultrasound, and a 3D ultrasound of the fetal face at approximately 20 weeks gestation identify fetuses with congenital anomalies and predict maternal and fetal complications?

DETAILED DESCRIPTION:
Pts will be consented upon presenting to the department for a comprehensive ultrasound.The 3D picture is the only part of the study that is not part of standard obstetrical care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at approximately 20 weeks
* ages 18-50
* singleton pregnancy
* plans to deliver at North Shore University Hosp
* completed step-wise sequential screening

Exclusion Criteria:

* multifetal gestation
* minors
* patients who have undergone diagnostic genetic testing
* incarcerated patients
* intention to deliver at a hospital other than North Shore University hosp

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women presenting for a comprehensive ultrasound at approximately 20 weeks
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2009-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Correlation of geometric morphometric analysis of fetal brow to 10 soft markers | completion of pregnancy
  In patients who have undergone step-wise sequential screening, how often will the evaluation of 10 midtrimester sonographic soft markers of aneuploidy such that the recommendation regarding invasive diagnostic testing be changed?

CONTACTS AND LOCATIONS:
Overall Officials: Burton Rochelson, MD, Principal Investigator — Northwell Health